CLINICAL TRIAL: NCT04380155
Title: Effects of Cycling Duration on Markers of Bone Metabolism in Active Young Men
Brief Title: Cycling Duration and Bone Markers in in Active Young Adults
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID restrictions all human studies have been suspended and not expected to resume. The PI decided to terminate the study.
Sponsor: Brock University (Other)
Collaborators: Natural Sciences and Engineering Research Council, Canada (Other)
Responsible Party: Principal Investigator, Panagiota Klentrou, Professor, Brock University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: REB 19-266
Record Dates: First submitted 2020-05-05; First posted 2020-05-08 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Bone Loss; Energy Supply; Deficiency
Keywords: Bone Turnover; biomarkers; cycling; energy availability; sclerostin; OPG/RANKL; bone formation; bone resorption
MeSH Terms: conditions — Bone Diseases, Metabolic; Sclerosteosis; Bone Resorption | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Single group, cross-over, random order
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants (Experimental): All participants will perform three moderate intensity cycling trials of different duration (30, 60 and 120 min) in an energy replete state.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Moderate intensity cycling trials of different duration (30, 60 and 120 min)

SUMMARY:
Exercise is an important factor in bone health. Sclerostin is one of the key molecules involved in bone response to mechanical loading. In particular, sclerostin decreases bone formation directly through the inhibition of Wnt/ β-catenin signaling and increases bone resorption indirectly via upregulation of the RANK/RANKL. The Wnt pathway is an anabolic signaling pathway, which leads to the activation of osteoblasts. OPG is another osteokine secreted by osteoblasts and osteogenic stomal cells that has a protective osteogenic role in humans by inhibiting the binding of RANKL to its receptor RANK. The RANK/RANKL pathway is a catabolic signaling pathway controlling osteoclast differentiation. Only a few studies have examined the effects of one single bout of high impact exercise on serum sclerostin levels in adults, most of which are from the investigators' lab. However, not many studies have examined the acute effects of moderate intensity, low-impact exercise on osteokines of the Wnt signaling. Previous studies have only investigated the impact of high intensity cycling on sclerostin, OPG and RANKL, however, no research has been done to investigate the response of osteokines to moderate intensity continuous cycling. This study aims to investigate differences in osteokines and markers of bone turnover following three moderate intensity cycling trials of different duration (30, 60 and 120 min) in an energy replete state. The question we aim to answer is whether there is a threshold of time where continued stimulus from moderate strain on the bone fails to elicit an additional metabolic response in bone or even becomes osteocatabolic, when athletes are in an energy replete state. Additional biochemical responses to the exercise will also be examined including inflammatory markers, glucose, anabolic/hormonal markers and oxidative stress.

DETAILED DESCRIPTION:
Introduction:

Exercise has been shown to positively benefit bone health. It's well documented that an acute bout of weight bearing, high load and dynamic strain on the skeleton mobilizes markers of bone formation in normal weight males and females. Acute bouts of low-impact high intensity exercise such as cycling, have also been investigated for their effects on bone formation and resorption, showing an overall anabolic effect (Mezil et al. 2015). One study exists investigating an acute two-hour bout of moderate intensity cycling, which showed increases in parathyroid hormone, associated with bone metabolism, although the effects of these transient hormonal changes on bone remain unknown (Barry & Kohrt, 2007). Minimal research has investigated the effects of acute bouts of moderate intensity continuous cycling (70% of VO2 max) on bone metabolism. In contrast to these acute controlled studies, at least two studies have reported that athletes who regularly participate in non-weight bearing sports such as cycling present with higher rates of osteopenia in the lumbar spine and hip region (Rector et al. 2008; Sherk et al. 2013). Another study investigated the bone status of adolescent male cyclists, over 17 and under 17 years of age, compared to healthy age matched controls. Cyclists had lower BMD at the legs, pelvis, and total hip. In cyclists over 17, reported BMD was 8.9% to 24.5% lower for the whole body, pelvis, femoral hip and legs, suggesting cycling performed during adolescent years may negatively affects bone health and one's ability to reach peak bone mass during this critical time (Olmedillas et al. 2011). However, a small study investigating 5 male elite racers during a 6-day road cycling stage race, while meeting energy needs, showed an increase markers of bone formation and a decrease in markers of bone resorption (Hinton et al. 2010). Thus, the evidence provided above appears contradictory. On the one hand, an acute bout of high intensity cycling has an osteogenic effect on bone, while longer-term studies or observational data, which allow for the time required to see changes in BMD, appear to show that road cycling can also have an osteocatabolic effect on bone (Olmedillas et al. 2012). This contradiction raises interesting questions about the impacts of larger loads of cycling, energy intakes, as well as the impacts of longer durations of cycling on bone health.

There appear to be conditions related to the sport of road cycling, not specific to the mechanics of cycling itself, that can predispose an athlete to low BMD over time. These conditions remain unclear. Possible factors contributing to the lower BMD found in cyclists include low energy availability and its associated hormonal and nutritional implications, carbohydrate availability, the omission of weight bearing loads due to long hours spent performing non-weight cycling, weight loss, as well as excess calcium losses through sweat and urine. Recent studies have also provided evidence of the importance of consuming carbohydrates in attenuating markers bone resorption and supporting bone health during exercise (Heikura et al. 2019). Of interest, is the fact that gymnasts, athletes who also often train under conditions of low energy availability, appear to gain a protective effect from their high impact sport, that overrides the bone resorption typically associated with calorie deficits. The high mechanical forces in this sport have large osteogenic effects, maintaining BMD, unlike what has been observed in cyclists (Robinson et al. 1995). This makes one question if it is the non-weight bearing nature of cycling, certain conditions surrounding cycling or something inherent to the mechanical aspects of cycling itself, that have a seemingly negative impact on bone?

To date, researchers have investigated the effects of an acute bout of high intensity cycling on markers of bone formation and resorption, as well as moderate intensity cycling and its effects on bone. Field studies have been executed where energy needs have been met and where energy deficiency was present. There is a gap in the research as far as the impact of duration of moderate intensity cycling on bone, in an energy replete state, in a controlled setting. Filling this gap through a systematic approach would help to better understand if and how duration impacts the metabolic bone response.

There are a variety of methods to measure the bone's response to acute mechanical loading. Since changes in BMD are not immediate, and only occur over longer time periods, this measurement is not appropriate to use to investigate changes in bone metabolism after one acute bout of exercise. After an acute bout of exercise, it is common to measure circulating bone turnover markers. These markers are products of bone formation or resorption. There are a variety of bone turnover markers, however some of the more commonly used are procollagen I intact N-terminal (PINP) and C-terminal crosslinking telopeptides of type I collagen (CTX), which are recognized by the International Osteoporosis Foundation (IOF) and are products of osteoblastic or osteoclastic cell activation, respectively. More recently, bone metabolism has been investigated through measures of the glycoprotein sclerostin, an inhibitor of the Wnt pathway, which leads to decreased bone formation. The Wnt/β-catenin signalling process has influence on the mobilization of OPG (Osteoprotegerin). OPG binds to receptor activator of nuclear factor kappa-β ligand (RANKL), preventing RANKL from binding to RANK (an osteoclast cell surface receptor), acting as a decoy receptor. RANKL binding to RANK would otherwise increase bone resorption. Therefore, the two pathways, Wnt-B-catenin and OPG/RANKL have a relationship that can help us to better understand the processes of bone resorption and formation.

Purpose: This study aims to investigate differences in markers of bone metabolism (CTX, PINP) and osteokines (sclerostin, OPG and RANKL) between three moderate intensity cycling trials of different duration (30, 60 and 120 min) in an energy and carbohydrate replete state. The question the investigators aim to answer is whether there is a threshold of time where continued stimulus from moderate strain on the bone fails to elicit an additional metabolic response in bone or even becomes osteocatabolic, when athletes are in an energy replete state. Additional biochemical responses to the exercise will also be examined including inflammatory markers, glucose, anabolic/hormonal markers and oxidative stress.

Methods:

Fifteen 20-30-year-old active male participants (sample size calculated based on Mezil et al. 2015) will arrive to the lab on 5 separate occasions. Visit one will include anthropometric measurements and a VO2max test. Participants will fill out a 24-hour food recall before visit one. Participants will complete one control and three continuous cycling trials (visits 2, 3, 4 and 5) on the cycle ergometer at 60-70% of their respective VO2 max based on their test from visit 1. The order of exercise sessions will be randomized.

Participants will follow a balanced diet the day before visits 2 to 5, which will be based on the participants food log for the 24 hours before visit one. Adjustments will be made to participants' food log in order to meet the macronutrient composition of 65% CHO, 25% PRO and 15% fat, to assure they arrive at the lab in an energy replete state before visits 2 to 5. Participants will also be given hydration guidelines for the 24 hours before arriving at the lab and will be asked to refrain from any vigorous activity for 24 hours before all visits to the lab.

For visits 2 to 5, participants will arrive at the lab fasted for a resting blood draw followed by a standard breakfast. Thirty minutes after breakfast, a post-breakfast blood draw will be taken followed by the respective protocol of the day (control, 30-, 60- or 120-min cycling). Additional blood samples will be taken as described below. To maintain hydration during the cycling trials, participants will be provided with 500 ml (for 30 min trial) to 1L (for the 60 and 120 min trials) of water to drink at libitum. The value of these visits is to see if there is a change in bone metabolism over time between the control, and three different cycling duration protocols.

Blood Samples: During the control session, a total of 7 blood samples will be taken: one upon arriving to the lab, one post-meal but before the 2-hour control session begins, and five during the control session at 30 min, 60 min, 120 min, 150 min and 180 min. During each cycling trial, a total of five (5) blood samples from each participant will be collected: one upon arriving to the lab, one post-meal but before cycling, and 3 post-cycling at 5 minutes, 30 minutes and 60 minutes after completion the cycling.

The blood samples will be drawn using a catheter (IV) performed by a certified paramedic. Catheterization would be upon subject arriving to the lab, suggest base line vital signs pre and post IV placement, preferably with subject in a recumbent position for the duration of assessment and IV placement. IV placement to be preferentially placed in the left or right forearm (posterior hand if no other sites visible) with a maximum of two IV attempts per visit. IV insertion to be completed using aseptic procedures as per safety standards. IV cannula to be secured via tegaderm, hypoallergenic tape and a compliant fishnet style elastic fabric to provide added protection from displacement during heavy perspiration and movement of the subject. Cannula would be locked with a saline lock and extension for access during blood draws (see below for schedule). Each blood draw should use one initial vacutainer as a waste draw due to saline in the IV lock with the second container being a pure venous sample. Once sampling is completed, saline is reintroduced at slightly higher pressure into the saline lock to maintain patency of the cannula for the next draw. Aseptic methods used throughout each procedure.

All blood samples will contain 5-10 ml of blood using serum and plasma tubes. Bone turnover markers, anabolic/hormonal markers, inflammatory markers and oxidative stress will be examined in each sample. To control for circadian rhythm, the exercise session and related blood samples will be performed at the same time of day between 9:00 am and 1:00pm.

Anthropometric Measurements: Height will be assessed using a stadiometer to the nearest 0.1 cm with no shoes. Body mass (kg), relative body fat (%) and fat free mass (kg) will be measured using Bod Pod (air displacement plethysmography method). All the participants will have familiarization with Bod Pod by sitting in the chamber before the test to see if they are claustrophobic. Participants will have the choice of an investigator of the same sex to take their anthropometric measurements.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian males,
* aged 20 to 30 years,
* healthy (not suffering from asthma),
* of normal weight (BMI: 18.5 - 25 kg/m2),
* recreationally active (i.e., regularly exercise 3-6 times per week, including 3 times of aerobic exercise over 45 min per session).

Exclusion Criteria:

* with no fracture over the last year,
* not taking any medication related to a chronic condition or bone health including food/nutritional supplements (e.g. protein, vitamin D, calcium),
* non-smokers,
* with no injuries or chronic conditions in which exercise may pose a risk (e.g., ACL or knee/hip/lower back injuries, arthritis, osteoporosis, neuromuscular diseases),
* currently not on a low carbohydrate or ketogenic diet.

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2023-10-29 (Actual); Study Completion 2023-10-29 (Actual)

PRIMARY OUTCOMES:
C-terminal crosslinking telopeptides of type I collagen (CTX) | 1 week
  Bone resorption marker (ng/ml)
Procollagen I intact N-terminal (PINP) | 1 week
  Bone formation marker (ng/ml)
Sclerostin (pg/ml) | 1 week
  Wnt related osteokine
Osteoprotegerin (OPG) | 1 week
  osteokine (pg/ml)
Receptor activator of nuclear factor kappa-β ligand (RANKL) | 1 week
  osteokine (pg/ml)

SECONDARY OUTCOMES:
Tumor necrosis factor alpha (TNF-a) | 1 week
  Pro-inflammatory cytokine (pg/ml)
Interleukin 10 (IL-10) | 1 week
  Anti-inflammatory cytokine (pg/ml)
Interleukin 6 (IL-6) | 1 week
  Myokine (pg/ml)
thiobarbituric acid reactive substances (TBARS) | 1 week
  oxidative stress marker
Glucose (ng/ml) | 1 week
  metabolic marker
Insulin growth factor one (IGF-1) | 1 week
  metabolic marker (ng/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Panagiota Klentrou, Principal Investigator — Brock University
Locations (1):
- Brock University, Saint Catharines, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mezil YA, Allison D, Kish K, Ditor D, Ward WE, Tsiani E, Klentrou P. Response of Bone Turnover Markers and Cytokines to High-Intensity Low-Impact Exercise. Med Sci Sports Exerc. 2015 Jul;47(7):1495-502. doi: 10.1249/MSS.0000000000000555. PMID 25373482
- [Background] Barry DW, Kohrt WM. Acute effects of 2 hours of moderate-intensity cycling on serum parathyroid hormone and calcium. Calcif Tissue Int. 2007 Jun;80(6):359-65. doi: 10.1007/s00223-007-9028-y. Epub 2007 Jun 5. PMID 17549534
- [Background] Sherk VD, Barry DW, Villalon KL, Hansen KC, Wolfe P, Kohrt WM. Bone loss over 1 year of training and competition in female cyclists. Clin J Sport Med. 2014 Jul;24(4):331-6. doi: 10.1097/JSM.0000000000000050. PMID 24326929
- [Background] Rector RS, Rogers R, Ruebel M, Hinton PS. Participation in road cycling vs running is associated with lower bone mineral density in men. Metabolism. 2008 Feb;57(2):226-32. doi: 10.1016/j.metabol.2007.09.005. PMID 18191053
- [Background] Olmedillas H, Gonzalez-Aguero A, Moreno LA, Casajus JA, Vicente-Rodriguez G. Bone related health status in adolescent cyclists. PLoS One. 2011;6(9):e24841. doi: 10.1371/journal.pone.0024841. Epub 2011 Sep 30. PMID 21980360
- [Background] Hinton PS, Rolleston A, Rehrer NJ, Hellemans IJ, Miller BF. Bone formation is increased to a greater extent than bone resorption during a cycling stage race. Appl Physiol Nutr Metab. 2010 Jun;35(3):344-9. doi: 10.1139/H10-025. PMID 20555379
- [Background] Heikura IA, Burke LM, Hawley JA, Ross ML, Garvican-Lewis L, Sharma AP, McKay AKA, Leckey JJ, Welvaert M, McCall L, Ackerman KE. A Short-Term Ketogenic Diet Impairs Markers of Bone Health in Response to Exercise. Front Endocrinol (Lausanne). 2020 Jan 21;10:880. doi: 10.3389/fendo.2019.00880. eCollection 2019. PMID 32038477
- [Background] Robinson TL, Snow-Harter C, Taaffe DR, Gillis D, Shaw J, Marcus R. Gymnasts exhibit higher bone mass than runners despite similar prevalence of amenorrhea and oligomenorrhea. J Bone Miner Res. 1995 Jan;10(1):26-35. doi: 10.1002/jbmr.5650100107. PMID 7747628